CLINICAL TRIAL: NCT03300206
Title: A Prospective, Block Stratified Clinical Trial to Evaluate the Performance and Operation of the Brevera Breast Biopsy System
Brief Title: A Post-Market Clinical Trial to Evaluate the Performance and Operation of the Brevera Breast Biopsy System
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-05B
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female
Keywords: Breast Biopsy; Breast Biopsy Imaging; Stereotactic Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Brevera Breast Biopsy System: The Brevera Breast Biopsy System with CorLumina imaging technology is a vacuum-assisted biopsy device, which is used to remove breast tissue in a minimally invasive manner using stereotactic or tomosynthesis imaging.
  Interventions: Device: Breast Biopsy
- Standard of Care: Each of the participating sites will currently be using a vacuum assisted breast biopsy system along with a specimen radiography system (or other specimen imaging system).
  Interventions: Device: Breast Biopsy

INTERVENTIONS:
Device: Breast Biopsy — A breast biopsy is a test that removes tissue or sometimes fluid from the suspicious area. The removed cells are examined under a microscope and further tested to check for the presence of breast cancer. A biopsy is a diagnostic procedure that can definitely determine if the suspicious area is cancerous.

SUMMARY:
The Brevera Breast Biopsy System integrates tissue acquisition, real time imaging, and post biopsy handling all during the same procedure. This post-market clinical trial will be performed to obtain clinical/operational data and feedback on the Brevera Breast Biopsy System as compared to the current standard-of-care breast biopsy procedures

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years of age or older
* Subject has at least one breast imaging finding requiring biopsy for which images are available
* Subject is able to understand, read and sign the trial specific informed consent form after the nature of the trial has been fully explained to her

Exclusion Criteria:

* Patients who, based on the physician's judgment, may be at increased risk or develop complications associated with core removal or biopsy.
* Patients receiving anticoagulant therapy or may have bleeding disorders which may put the patient at increased risk of procedural complications based upon physicians judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females (biologic) will be eligible for participation in the clinical trial.
Study Population: Female subjects who require a stereotactic breast biopsy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - HonorHealth, Phoenix, Arizona
  - Kensington Medical Center - Kaiser Permanente, Kensington, Maryland
  - Washington University, St Louis, Missouri
  - Elizabeth Wende Breast Center, Rochester, New York
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brevera Breast Biopsy System | Standard of Care
Started | 316 | 209
Completed | 316 | 209
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brevera Breast Biopsy System | Standard of Care | Total
Number analyzed (Participants) | 316 | 209 | 525
Age, Customized [Mean (Standard Deviation); unit: years] | 57.80 (11.25) | 58.08 (11.93) | 57.91 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 209 | 525
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference in Procedural Time in Minutes
Description: The primary endpoint of this trial is the measured difference in procedure time between biopsies performed with the Brevera biopsy system and those performed with the standard-of-care biopsy systems at each clinical site. Additionally, feedback from the perspective of the participant radiologists, technologists, and subjects using the systems was reported.
Time Frame: Average Time- Procedure (1 Lesion per subject): Total Time elapsed from when the subject enters the procedure room until they have left the procedure room, an average of 43 minutes.
Population: This study involved the participation of 525 female patients aged 18 years or older with suspicious findings on mammographic screening or diagnostic exams who were sent for breast biopsy. These subjects were enrolled at seven different clinical sites (75 subjects per site) and then separated to have their biopsy procedure performed using the current standard of care breast biopsy procedure (209) or the Brevera Breast Biopsy system (316).
Measure: Mean (Standard Deviation); unit: procedure time in minutes
Arm/Group | Brevera Breast Biopsy System | Standard of Care
Number analyzed (Participants) | 316 | 209
procedure time in minutes | 42.15 (14.06) | 40.13 (12.14)

2. Secondary Outcome: Post-biopsy Complication Rates
Description: Adverse event percentage rates.
Time Frame: The time of consent until the subject procedure was completed, an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Brevera Breast Biopsy System | Standard of Care
Number analyzed (Participants) | 316 | 209
Participants | 9 | 4

3. Secondary Outcome: Number of Samples Collected Per Lesion
Description: Number of samples collected per lesion
Time Frame: Samples collected from day of Breast Biopsy Procedure Only
Measure: Mean (Standard Deviation); unit: samples obtained
Arm/Group | Brevera Breast Biopsy System | Standard of Care
Number analyzed (Participants) | 265 | 159
samples obtained | 6.69 (3.39) | 7.25 (2.69)

4. Secondary Outcome: Percentage of Procedures With Overall Positive Opinion From Radiologists, Technologists and Patients
Description: The radiologists, technologists, and patients participating in this study were asked to provide feedback on the Brevera Biopsy System at the completion of each procedure. Their responses (raw scores) were reported and converted to percentage of procedures with overall positive opinion. The scale goes from 0% (poor/negative opinion) to 100% (excellent/positive opinion).
Time Frame: Through study completion, enrollment expected to take up to 6-10 months at each participant site. Data collected from day of Breast Biopsy Procedure Only
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Groups:
- Radiologist Feedback: Radiologist with a positive overall opinion of the Brevera Breast Biopsy System for the procedure (scored 3, 4 or 5 on Likert Scale).
- Technologist Feedback: Technologist with a positive overall opinion of the Brevera Breast Biopsy System for procedures (scored 3, 4 or 5 on Likert Scale).
- Subject Feedback: Subjects agreed that they were satisfied with the facility and the care that they received during the procedure (scored 3, 4 or 5 on Likert Scale).
Arm/Group | Radiologist Feedback | Technologist Feedback | Subject Feedback
Number analyzed (Participants) | 301 | 301 | 296
percentage of procedures | 79.8 [8.9 to 91.1] | 72.8 [6.6 to 94.4] | 99.0 [0.3 to 99.7]

ADVERSE EVENTS:
Time Frame: 2 hours: per the standard of care protocol, each subject participating in this study was evaluated for any adverse events from the time the biopsy procedure began to the time the subject was released from the outpatient treatment facility.
Description: No serious adverse events were reported in this study.
Arm/Group | Brevera Breast Biopsy System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/316 | 0/209
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/209
Other Adverse Events (participants affected / at risk) | 9/316 | 4/209
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brevera Breast Biopsy System (N=316) | Standard of Care (N=209)
Anticipated Adverse Events (Injury, poisoning and procedural complications) | 9 (9) | 4 (4) — Most of the observed anticipated adverse events were related to syncope/fainting/panic attack/excessive bleeding (1 case)/hematoma (1 case). All these events were resolved the same day they started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication by the collaborative participants is not being conceived or submitted within 10 months following the conclusion of enrollment at the last enrolling site, an individual site may petition to publish his or her site data independently of the group. Hologic will advise on the status of publications in process and determine when individual results may be released.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03300206/Prot_SAP_000.pdf